CLINICAL TRIAL: NCT00995605
Title: AMAP102 - A Phase I, Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetics Study in Healthy Subjects
Brief Title: AMAP102 - Safety, Tolerability and Pharmacokinetics in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Reached sufficient pharmacokinetic exposures
Sponsor: AnaMar AB (Industry)
Responsible Party: Clinical Manager
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102-240-01; 2008-004940-35; 2704-026
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Groups SAD (Experimental): AMAP102 or Placebo as single ascending doses in five groups
  Interventions: Drug: AMAP102
- Groups MAD (Experimental): AMAP102 or Placebo as multiple ascending doses twice daily for seven days in two groups
  Interventions: Drug: AMAP102

INTERVENTIONS:
Drug: AMAP102 — AMAP102 or Placebo

SUMMARY:
The purpose of this study is to determine whether AMAP102 is safe and well tolerated by humans.

ELIGIBILITY:
Inclusion Criteria:

1. In Groups A, B, D, E and F, subjects will be males of any ethnic origin between 18 and 65 years of with a BMI between 20.0 and 30.0 kg/m2
2. In Group C, subjects will be females (of non-childbearing potential) of any ethnic origin between 18 and 65 years with a BMI between 20.0 and 28.0 kg/m2
3. For Group C, women will be of non-childbearing potential, defined as surgically sterile or post-menopausal, non-lactating and having a negative serum pregnancy test
4. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead ECG and clinical laboratory evaluations
5. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

1. Male subjects who are not willing to use appropriate contraception from the time of the first dose until 3 months after the final dosing occasion
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration
3. Subjects who have used any non-prescribed systemic or topical medication within 7 days of the first dose administration
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration
5. Subjects who are still participating in a clinical study or who have participated in a clinical study involving administration of an investigational drug in the past 3 months
6. Subjects who have donated any blood, plasma or platelets in the month prior to screening or who have made donations on more than two occasions within the 12 months preceding the first dose administration
7. Subjects with a significant history of drug allergy as determined by the Investigator
8. Subjects who have any clinically significant allergic disease as determined by the Investigator
9. Subjects who have a supine blood pressure and supine pulse rate higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 40 bpm, respectively
10. Subjects who consume more than 28 units (males) or more than 21 units (females) of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits)
11. Subjects who smoke more than 10 cigarettes or the equivalent in tobacco per day
12. Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorders as determined by the Investigator
13. Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator
14. Subjects who are known to have serum hepatitis, or who are carriers of the HBsAg or hepatitis C antibody, or who have a positive result to the test for HIV antibodies
15. Subjects who have an abnormality in the 12-lead ECG such that, in the opinion of the investigator, increases the risk of participating in the study, such as QTc(b) interval greater than 430 msec (male) or greater than 450 msec (female), 2nd or 3rd degree Atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as PR shorter than 110 msec, confirmed by a repeat ECG
16. Subjects with a significant cardiac history (e.g. heart failure, hypokalemia, long QT syndrome), significant history of fainting, syncope or family history of sudden cardiac death
17. Subjects who, in the opinion of the Investigator, should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability determined by adverse events, vital signs, ECG and clinical laboratory evaluations | During residential period and at follow up visit

SECONDARY OUTCOMES:
Investigate the pharmacokinetic profile of AMAP102 after one oral dose and after multiple oral doses during twice daily dosing for seven days, and compare the pharmacokinetic profile for men and women | PK sampling at defined timepoints during residential period

CONTACTS AND LOCATIONS:
Overall Officials: Dr Joseph Chiesa, MD FFPM FICR CSci, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom